CLINICAL TRIAL: NCT04901351
Title: Feasibility of a Multi-site Screening Strategy in HPV+ Patients at High Risk of Cancer, With Characterization of the HPV Subtypes Involved by High Throughput Sequencing Technique: DEP-HPV
Brief Title: Multi-site HPV Screening by High-throughput Sequencing in Patients With Chronic HPV-HR Infection Followed by Gynecology
Acronym: DEP-HPV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/21/0009
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Human Papillomavirus
Keywords: Cervical cancer; Anal cancer;; ENT cancer; Next generation sequencing
MeSH Terms: conditions — Uterine Cervical Neoplasms; Anus Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients chronically infected with HPV (Experimental): The study will be offered to patients with chronic HPV infection as part of an annual consultation scheduled in the gynecology care package.
  Interventions: Procedure: Smear

INTERVENTIONS:
Procedure: Smear — In addition to the routine gynecological follow-up including a cervico-vaginal smear and an HPV test (HPV-HR genome detection), the doctor will propose prospectively to all consecutive patients who meet the inclusion criteria, during a follow-up consultation (post treatment of cervical dysplasia), to participate in the study, that is to have 2 other anal and ENT samples for an HPV test

SUMMARY:
The main risk of developing cervical cancer is the persistence of an High risk human papillomavirus (HPV-HR) infection, the mechanisms of which are still not understood. These chronically infected patients could develop multi-site lesions. The main objective is to assess the feasibility of setting up a personalized screening in patients at high risk of cervical cancer (chronically infected with HPV), by evaluating documenting the acceptability of these patients to be sampled from the ENT sphere and anal spheres for HPV analysis with next-generation sequencing.

DETAILED DESCRIPTION:
Screening for cervical cancer (CCU) is based on a well-codified, organized national screening program. However, unlike breast cancer or colorectal cancer, there is no personalized screening for patients said identified to be at higher risk of developing UCC. In addition, other cancers linked to HPV (papillomavirus), oropharynx and anal, were excluded from this screening, including for high-risk patients. However, in France, HPV-related cancers in the majority of cases concern the cervix (44%), but the anal (24%) and oropharynx (22%) locations can no longer be neglected. An increase of more than 200% in the incidence of oropharyngeal cancer was reported in the United States between 1988 and 2004. There appears to be a significant association between certain some sexual habits and the risk of multi-site HPV (+) carcinoma. However, several studies suggested that multi-site transmission could involve simple self-inoculation. Therefore, the investigators are interested in a population particularly at risk of developing these viro-induced cancers: patients chronically infected with HPV who will also be those likely to develop multi-site lesions. It is established that high risk HPV are more widely involved in CCU, however, the causes of the persistence of these HPV have not been clearly identified.

It therefore seems essential to continue screening for CCU in chronically infected patients, taking into account the multiple possible locations. The characterization of HPV viruses in terms of types, subtypes and co-infections is one of the key elements, determining the risk of persistence and the risk of cancer. Also, the implementation of a multi-site screening associated with a genotyping by high throughput or new generation sequencing (NGS) would make it possible to understand the part of HPV in the persistence of the infection and to detect the development of lesions at other anatomical sites.

ELIGIBILITY:
Inclusion Criteria:

-Chronic infected patients defined by: Patients with persistent HPV-HR cytological infection (high risk) (as early as 6 months post-treatment of a cervical or vaginal injury), or a recurrence of a high-grade squamous intraepithelial lesion (CIN2 or CIN3 or HSIL) or a recurrence of cancer in the cervix or vagina

* Patients who have given their written consent to participate in the study.
* Person affiliated or beneficiary of a social security scheme.

Exclusion Criteria:

Patient with an infection or a persistent lesion after treatment or not, linked only to low-risk HPV.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Acceptance by the patient (yes / no binary variable) of ENT and / or anal samples in addition to the cervical sample during an annual gynecological follow-up. | Inclusion day (day 0)
Number of sites sampled | Inclusion day (day 0)
  It will be collected anonymously if spontaneously explained by the patient.
Reasons for refusing multi-site samples | Inclusion day (day 0)

SECONDARY OUTCOMES:
Positivity to HPV tests for at least one of the other sites (ENT or anal) | Inclusion day (day 0)
Identification of HPV + subtypes on the different sites | Inclusion day (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Elodie Chantalat, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No